CLINICAL TRIAL: NCT00614939
Title: A Short-term 12-Week, Multi-centre, Randomized, Parallel-group, Double-blind, Placebo-controlled Study to Evaluate the Treatment Effect of Saxagliptin Compared With Placebo in Adult Patients With Type 2 Diabetes and Renal Impairment (Moderate, Severe, and End-Stage) With an Additional 40-week, Randomized, Double-blind, Placebo-controlled Long-term Observational Period.
Brief Title: Treatment Effect of Saxagliptin Compared With Placebo in Patients With Type 2 Diabetes and Renal Impairment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Peter Ohman, MD, PhD, Medical Science Director, AstraZeneca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1680C00007; EudraCT number 2007-004951-12
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2010-07-07 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Type 2 Diabetes
Keywords: DPP-4 inhibitors; HbA1c; incretins; Renal Impairment
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency | interventions — saxagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saxa (Experimental): Saxagliptin
  Interventions: Drug: Saxagliptin
- Placebo (No Intervention): Placebo to match
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Saxagliptin — 2.5 mg once daily oral dose
  Other Names: Onglyza
  Arms: Saxa
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Saxagliptin is a new investigational medication being developed for treatment of type 2 diabetes. This study is designed to test the efficacy of once daily saxagliptin in renally impaired patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes
* Documented history of CrCl <50 ml/min within the 3 months prior to enrollment
* HbA1c ≥7.0% and ≤11.0%

Exclusion Criteria:

* Type 1 diabetes, history of diabetic ketoacidosis or hyposmolar non-ketonic coma
* Previous or current treatment with any DPP-IV inhibitor and/or GLP-1 mimetic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2008-01; Primary Completion 2009-06 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ohman, MD, PhD, Study Director — AstraZeneca; Deborah Price, MSc, Study Chair — AstraZeneca
Locations (74):
- United States (11):
  - Research Site, Concord, California
  - Research Site, Sacramento, California
  - Research Site, Denver, Colorado
  - Research Site, Topeka, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Great Falls, Montana
  - Research Site, Greenville, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Corpus Christi, Texas
  - Research Site, Charleston, West Virginia
- Belarus (3):
  - Research Site, Brest
  - Research Site, Homyel
  - Research Site, Minsk
- Bulgaria (3):
  - Research Site, Dimitrovgrad
  - Research Site, Sofia
  - Research Site, Veliko Tarnovo
- Croatia (5):
  - Research Site, Rijeka, Croatia
  - Research Site, Karlovac
  - Research Site, Osijek
  - Research Site, Split
  - Research Site, Zagreb
- Czechia (5):
  - Research Site, Moravský Krumlov
  - Research Site, Prague
  - Research Site, Teplice
  - Research Site, Ústí nad Labem
  - Research Site, Znojmo
- Research Site, Tallinn, Estonia
- Germany (5):
  - Research Site, Dieburg
  - Research Site, Düsseldorf
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Mannheim
- Hungary (5):
  - Research Site, Debrecen
  - Research Site, Győr
  - Research Site, Kalocsa
  - Research Site, Kecskemét
  - Research Site, Zalaegerszeg
- Research Site, Riga, Latvia
- Lithuania (4):
  - Research Site, Kaunas
  - Research Site, Klaipėda
  - Research Site, Panevezys
  - Research Site, Vilnius
- Poland (13):
  - Research Site, Lodz, 90-153
  - Research Site, Bialystok
  - Research Site, Ciechanów
  - Research Site, Golub-Dobrzyń
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Katowice
  - Research Site, Krakow
  - Research Site, Maków Mazowiecki
  - Research Site, Radom
  - Research Site, Szczecin
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zabrze
- Romania (5):
  - Research Site, Bacau, Bacău
  - Research Site, Brasov, Brașov County
  - Research Site, Satu Mare, Satu Mare County
  - Research Site, Bucharest
  - Research Site, Sf Gheorghe
- Russia (5):
  - Research Site, Chelyabinsk
  - Research Site, Moscow
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Yaroslavl
- Ukraine (8):
  - Research Site, Dnipropetrovsk
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Mykolayiv
  - Research Site, Sumy
  - Research Site, Ternopil
  - Research Site, Zaporizhzhya

REFERENCES:
- [Derived] Nowicki M, Rychlik I, Haller H, Warren ML, Suchower L, Gause-Nilsson I; D1680C00007 Investigators. Saxagliptin improves glycaemic control and is well tolerated in patients with type 2 diabetes mellitus and renal impairment. Diabetes Obes Metab. 2011 Jun;13(6):523-32. doi: 10.1111/j.1463-1326.2011.01382.x. PMID 21332627

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 572 participants were enrolled in the study; 561 entered the Lead-in period and 170 patients were randomized and treated.
Groups:
- Saxa: Saxagliptin 2.5 mg once daily oral dose
Period: Overall Study
Arm/Group | Placebo | Saxa
Started | 85 (Randomized and treated) | 85 (Randomized and treated)
Completed | 50 (Completed 52 weeks of treatment) | 42 (Completed 52 weeks of treatment)
Not Completed | 35 | 43
Not completed — Withdrawal by Subject | 10 | 17
Not completed — Study specific discontinuation criteris | 13 | 16
Not completed — Adverse Event | 2 | 5
Not completed — Incorrect enrollment | 1 | 2
Not completed — Death | 4 | 3
Not completed — Poor/non-compliance | 4 | 0
Not completed — Hospitalized due to kidney transplant | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Saxa | Total
Number analyzed (Participants) | 85 | 85 | 170
Age Continuous [Mean (Standard Deviation); unit: years] | 66.2 (9.08) | 66.8 (8.27) | 66.5 (8.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 53 | 97
  Male | 41 | 32 | 73
Baseline Renal Impairment Category [Number; unit: Participants]
  Moderate | 42 | 48 | 90
  Severe | 23 | 18 | 41
  End-Stage | 20 | 19 | 39
Baseline Diabetes Therapy [Number; unit: participants]
  Diabetes Therapy | 84 | 83 | 167
  Insulin | 57 | 71 | 128
  Oral blood glucose lowering drug | 30 | 23 | 53

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Glycosylated Haemoglobin A1c (HbA1c) Level to Week 12 Last Observation Carried Forward (LOCF)
Description: Adjusted* mean change from baseline in HbA1c achieved with saxagliptin 2.5 mg once daily versus placebo at Week 12 (Full Analysis Set). HbA1c is a continuous measure, the change from baseline for each participant is calculated at the Week 12 value minus the baseline value.
Time Frame: Baseline , Week 12 (LOCF)
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis: change from baseline to Week 12 (LOCF) for efficacy, subjects must have had a baseline and at least 1 post-baseline efficacy measurement.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Saxa
Number analyzed (Participants) | 83 | 81
Percent
  Baseline | 8.09 (0.119) | 8.45 (0.135)
  Week 12 | 7.80 (0.137) | 7.63 (0.132)
  Adjusted Mean Change from Baseline | -0.44 (0.109) | -0.86 (0.112)
Statistical Analysis 1: Comparison: Placebo vs Saxa; Test type: Superiority or Other; p = 0.007, ANCOVA; *Adjusted for baseline HbA1c; Mean Difference (Net) = -0.42, 95% CI 2-sided [-0.71 to -0.12], Standard Error of Mean 0.151

2. Secondary Outcome: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) to Week 12 (LOCF)- Moderate Renal Impairment Subgroup
Description: Adjusted* mean change from baseline in fasting plasma glucose (FPG) achieved with saxagliptin 2.5 mg once daily versus placebo at Week 12 (Full Analysis Set) for the moderate renal impairment subgroup. FPG is a continuous measure, the change from baseline for each participant is calculated at the Week 12 value minus the baseline value.
Time Frame: Baseline, Week 12 (LOCF)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Saxa
Number analyzed (Participants) | 40 | 44
mg/dL
  Baseline | 162.33 (8.933) | 202.82 (9.858)
  Week 12 | 174.50 (10.089) | 173.91 (7.938)
  Adjusted Mean Change from Baseline | -2.88 (9.073) | -15.22 (8.630)
Statistical Analysis 1: Comparison: Placebo vs Saxa; Additional details about the analysis, such as null hypothesis and power calculation: Due to a statistically significant treatment-by-baseline renal impairment interaction, fasting plasma glucose results were analyzed separately for each baseline renal impairment category; Test type: Superiority or Other; p = 0.339, ANCOVA; *Adjusted for baseline FPG; Mean Difference (Net) = -12.34, 95% CI [-37.91 to 13.22], Standard Error of Mean 12.847

3. Secondary Outcome: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) to Week 12 (LOCF) - Severe Renal Impairment Subgroup
Description: Adjusted* mean change from baseline in fasting plasma glucose (FPG) achieved with saxagliptin 2.5 mg once daily versus placebo at Week 12 (Full Analysis Set) for the severe renal impairment subgroup. FPG is a continuous measure, the change from baseline for each participant is calculated at the Week 12 value minus the baseline value.
Time Frame: Baseline, Week 12 (LOCF)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Saxa
Number analyzed (Participants) | 23 | 18
mg/dL
  Baseline | 173.48 (11.630) | 165.50 (19.909)
  Week 12 | 141.52 (14.276) | 133.83 (11.371)
  Adjusted mean change | -29.91 (11.212) | -34.28 (12.677)
Statistical Analysis 1: Comparison: Placebo vs Saxa; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.798, ANCOVA; *Adjusted for baseline FPG; Mean Difference (Net) = -4.36, 95% CI 2-sided [-38.65 to 29.93], Standard Error of Mean 16.938

4. Secondary Outcome: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) to Week 12 (LOCF) - End-Stage Renal Impairment Subgroup
Description: Adjusted* mean change from baseline in fasting plasma glucose (FPG) achieved with saxagliptin 2.5 mg once daily versus placebo at Week 12 (Full Analysis Set) for the end-stage renal impairment subgroup. FPG is a continuous measure, the change from baseline for each participant is calculated at the Week 12 value minus the baseline value.
Time Frame: Baseline, Week 12 (LOCF)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Saxa
Number analyzed (Participants) | 18 | 15
mg/dL
  Baseline | 170.39 (14.518) | 177.07 (10.638)
  Week 12 | 161.11 (12.624) | 207.60 (30.515)
  Adjusted mean change | -11.18 (20.752) | 32.82 (22.737)
Statistical Analysis 1: Comparison: Placebo vs Saxa; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.164, ANCOVA; *Adjusted for baseline FPG; Mean Difference (Net) = 44.01, 95% CI 2-sided [-18.93 to 106.94], Standard Error of Mean 30.815

5. Secondary Outcome: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) to Week 12 (LOCF) - Moderate Renal Impairment Subgroup
Description: as for outcome 2
Time Frame: Baseline, Week 12 (LOCF)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Saxa
Number analyzed (Participants) | 40 | 44
mmol/L
  Baseline | 9.01 (0.495) | 11.25 (0.548)
  Week 12 | 9.68 (0.560) | 9.65 (0.441)
  Absolute mean change | -0.16 (0.504) | -0.84 (0.479)
Statistical Analysis 1: Comparison: Placebo vs Saxa; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Footnote; *Adjusted for baseline FPG; Mean Difference (Net) = -0.68, 95% CI 2-sided [-2.10 to 0.74], Standard Error of Mean 0.713

6. Secondary Outcome: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) to Week 12 (LOCF) - Severe Renal Impairment Subgroup
Description: as for outcome 3
Time Frame: Baseline, Week 12 (LOCF)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Saxa
Number analyzed (Participants) | 23 | 18
mmol/L
  Baseline | 9.63 (0.646) | 9.17 (1.105)
  Week 12 | 7.86 (0.793) | 7.43 (0.632)
  Adjusted mean change | -1.66 (0.623) | -1.89 (0.704)
Statistical Analysis 1: Comparison: Placebo vs Saxa; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Footnote; *Adjusted for baseline FPG; Mean Difference (Net) = -0.24, 95% CI 2-sided [-2.14 to 1.67], Standard Error of Mean 0.941

7. Secondary Outcome: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) to Week 12 (LOCF) - End-Stage Renal Impairment Subgroup
Description: as for outcome 4
Time Frame: Baseline, Week 12 (LOCF)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Saxa
Number analyzed (Participants) | 18 | 15
mmol/L
  Baseline | 9.46 (0.807) | 9.83 (0.591)
  Week 12 | 8.94 (0.700) | 11.52 (1.692)
  Adjusted mean change | -0.62 (1.151) | 1.81 (1.261)
Statistical Analysis 1: Comparison: Placebo vs Saxa; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Footnote; *Adjusted for baseline FPG; Mean Difference (Net) = 2.44, 95% CI 2-sided [-1.05 to 5.93], Standard Error of Mean 1.709

8. Secondary Outcome: Absolute Change From Baseline in Glycosylated Haemoglobin A1c (HbA1c) Level to Week 52
Description: Adjusted* mean change from baseline in HbA1c achieved with saxagliptin 2.5 mg once daily versus placebo at Week 52 (Full Analysis Set). HbA1c is a continuous measure, the change from baseline for each participant is calculated at the Week 52 value minus the baseline value.
Time Frame: Baseline , Week 52
Population: Randomized participants who took at least 1 dose of double-blind treatment. To be included in analysis: change from baseline to Week 52 for efficacy, subjects must have had a baseline and at least 1 post-baseline efficacy measurement. Data were excluded after changes in oral blood glucose lowering drug or insulin.
Measure: Mean (Standard Error); unit: Percent
Arm/Group | Placebo | Saxa
Number analyzed (Participants) | 82 | 78
Percent
  Baseline | 8.10 (0.120) | 8.44 (0.134)
  Week 52 | 7.93 (0.173) | 7.41 (0.138)
  Adjusted mean change | -0.53 (0.154) | -1.35 (0.174)
Statistical Analysis 1: Comparison: Placebo vs Saxa; Test type: Superiority or Other; Repeated Measures; Number of subjects with observed values at Week 52 was n=26 for saxagliptin and n=34 for placebo *Adjusted for baseline HbA1c; Mean Difference (Net) = -0.82, 95% CI 2-sided [-1.27 to -0.37], Standard Error of Mean 0.228

9. Secondary Outcome: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) to Week 52 - Moderate Renal Impairment Subgroup
Description: Adjusted* mean change from baseline in fasting plasma glucose (FPG) achieved with saxagliptin 2.5 mg once daily versus placebo at Week 52 (Full Analysis Set) for the moderate renal impairment subgroup. FPG is a continuous measure, the change from baseline for each participant is calculated at the Week 52 value minus the baseline value.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Saxa
Number analyzed (Participants) | 40 | 44
mg/dL
  Baseline | 162.33 (8.933) | 202.82 (9.858)
  Week 52 | 174.83 (11.295) | 177.43 (7.637)
  Adjusted mean change | 3.02 (13.277) | -14.96 (12.873)
Statistical Analysis 1: Comparison: Placebo vs Saxa; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Repeated Measures; Number of subjects with observed values at Week 52 was n=17 for saxagliptin and n=16 for placebo *Adjusted for baseline FPG; Mean Difference (Net) = -17.98, 95% CI 2-sided [-54.28 to 18.33], Standard Error of Mean 18.475

10. Secondary Outcome: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) to Week 52 - Severe Renal Impairment Subgroup
Description: Adjusted* mean change from baseline in fasting plasma glucose (FPG) achieved with saxagliptin 2.5 mg once daily versus placebo at Week 52 (Full Analysis Set) for the severe renal impairment subgroup. FPG is a continuous measure, the change from baseline for each participant is calculated at the Week 52 value minus the baseline value.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Saxa
Number analyzed (Participants) | 23 | 18
mg/dL
  Baseline | 173.48 (11.630) | 165.50 (19.909)
  Week 52 | 151.78 (9.896) | 139.06 (12.408)
  Adjusted mean change | -24.59 (14.510) | -40.32 (20.789)
Statistical Analysis 1: Comparison: Placebo vs Saxa; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Repeated Measures; Number of subjects with observed values at Week 52 was n=5 for saxagliptin and n=11 for placebo. *Adjusted for baseline FPG; Mean Difference (Net) = -15.73, 95% CI 2-sided [-65.77 to 34.30], Standard Error of Mean 25.326

11. Secondary Outcome: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) to Week 52 - End-Stage Renal Impairment Subgroup
Description: Adjusted* mean change from baseline in fasting plasma glucose (FPG) achieved with saxagliptin 2.5 mg once daily versus placebo at Week 52 (Full Analysis Set) for the end-stage renal impairment subgroup. FPG is a continuous measure, the change from baseline for each participant is calculated at the Week 52 value minus the baseline value.
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Saxa
Number analyzed (Participants) | 18 | 15
mg/dL
  Baseline | 170.39 (14.518) | 177.07 (10.638)
  Week 52 | 161.94 (13.097) | 214.27 (31.740)
  Adjusted mean change | -2.18 (29.226) | -40.28 (45.470)
Statistical Analysis 1: Comparison: Placebo vs Saxa; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Repeated Measures; Number of subjects with observed values at Week 52 was n=2 for saxagliptin and n=5 for placebo. *Adjusted for baseline FPG; Mean Difference (Net) = -38.09, 95% CI 2-sided [-144.44 to 68.26], Standard Error of Mean 53.822

12. Secondary Outcome: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) to Week 52 - Moderate Renal Impairment Subgroup
Description: as for outcome 9
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Saxa
Number analyzed (Participants) | 40 | 44
mmol/L
  Baseline | 9.01 (0.495) | 11.25 (0.548)
  Week 52 | 9.70 (0.627) | 9.85 (0.424)
  Adjusted mean change | 0.15 (0.738) | -0.82 (0.715)
Statistical Analysis 1: Comparison: Placebo vs Saxa; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Repeated Measures; Number of subjects with observed values at Week 52 was n=17 for saxagliptin and n=16 for placebo. *Adjusted for baseline FPG; Mean Difference (Net) = -0.97, 95% CI 2-sided [-2.99 to 1.04], Standard Error of Mean 1.027

13. Secondary Outcome: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) to Week 52 - Severe Renal Impairment Subgroup
Description: as for outcome 10
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Saxa
Number analyzed (Participants) | 23 | 18
mmol/L
  Baseline | 9.63 (0.646) | 9.17 (1.105)
  Week 52 | 8.42 (0.551) | 7.71 (0.688)
  Adjusted mean change | -1.37 (0.805) | -2.25 (1.154)
Statistical Analysis 1: Comparison: Placebo vs Saxa; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Repeated Measures; [statistical method as in outcome 10, analysis 1]; Mean Difference (Net) = -0.89, 95% CI 2-sided [-3.66 to 1.89], Standard Error of Mean 1.405

14. Secondary Outcome: Absolute Change From Baseline in Fasting Plasma Glucose (FPG) to Week 52 - End-Stage Renal Impairment Subgroup
Description: as for outcome 11
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Placebo | Saxa
Number analyzed (Participants) | 18 | 15
mmol/L
  Baseline | 9.46 (0.807) | 9.83 (0.591)
  Week 52 | 8.99 (0.728) | 11.89 (1.760)
  Adjusted mean change | -0.11 (1.621) | -2.25 (2.522)
Statistical Analysis 1: Comparison: Placebo vs Saxa; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Repeated Measures; [statistical method as in outcome 11, analysis 1]; Mean Difference (Net) = -2.14, 95% CI 2-sided [-8.04 to 3.76], Standard Error of Mean 2.985

ADVERSE EVENTS:
Arm/Group | Placebo | Saxa
Serious Adverse Events (participants affected / at risk) | 24/85 | 23/85
Other Adverse Events (participants affected / at risk) | 36/85 | 38/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=85) | Saxa (N=85)
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 2
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Pyelonephritis Acute (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Poor Peripheral Circulation (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 1 | 0
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1
Alanine Aminotransferase Increased (Investigations) | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Malignant Fibrous Histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 1 | 1
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Pneumonia (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 0 | 1
Infected Skin Ulcer (Infections and infestations) | 1 | 0
Lobar Pneumonia (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Bifascicular Block (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 2 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Cauda Equina Syndrome (Nervous system disorders) | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1
Cerebral Hypoperfusion (Nervous system disorders) | 1 | 0
Arteriovenous Fistula (Vascular disorders) | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 1 | 0
Femoral Artery Occlusion (Vascular disorders) | 1 | 0
Peripheral Ischaemia (Vascular disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Iridocyclitis (Eye disorders) | 0 | 1
Pseudoexfoliation Of Lens Capsule (Eye disorders) | 0 | 1
Sudden Death (General disorders) | 2 | 1
Oedema (Gastrointestinal disorders) | 1 | 0
Blood Glucose Increased (Investigations) | 0 | 1
Calculus Ureteric (Renal and urinary disorders) | 0 | 1
Renal Failure Chronic (Renal and urinary disorders) | 1 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Arteriovenous Fistula Thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arteriovenous Fistula Operation (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=85) | Saxa (N=85)
Hypoglycaemia (Metabolism and nutrition disorders) | 25 | 24
Anaemia (Blood and lymphatic system disorders) | 7 | 5
Oedema Peripheral (General disorders) | 6 | 2
Urinary Tract Infection (Infections and infestations) | 3 | 5
Hypertension (Vascular disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No